CLINICAL TRIAL: NCT06841419
Title: Reliability and Versatility of Pedicled Anterolateral Thigh Flap in Reconstruction of Soft Tissue Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abdelnasser Mohamed Ahmed, Resident in Plastic Surgery Department Suhag university, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med--12-1-03MS
Record Dates: First submitted 2025-01-24; First posted 2025-02-24 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Post Traumatic Soft Tissue Defects That Could be Reached by Pedicled Anterolateral Thigh Flap; Post Tumor Excision Soft Tissue Defects; Post Debridement Soft Tissue Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- a group of patients with hip, thighs, knees and lower abdomen regions soft tissue defects (Experimental): treating patients of the group mentioned by reconstructing their tissue defects by pedicled anterolateral thigh flap.
  Interventions: Procedure: surgical reconstruction of a soft tissue defects by a pedicled flap

INTERVENTIONS:
Procedure: surgical reconstruction of a soft tissue defects by a pedicled flap — harvesting of a fasciocutaneous flap from the anterolateral aspect of thigh based on a perforators from the descending branch of lateral femoral circumflex artery to reconstruct a neighboring soft tissue defect.

SUMMARY:
a prospective case series study for evaluation of the reliability and versatility of pedicled anterolateral thigh flap in the reconstruction of soft tissue defects as regards flap survival and complications, donor site morbidity and aesthetic outcome.

ELIGIBILITY:
Inclusion Criteria:

* All patients with clean hip, thighs or lower abdomen defects either traumatic or non_traumatic that cannot be closed primarily.

Exclusion Criteria:

* Patients with possible compromise of vascular pedicle due to previous trauma or surgery.
* Patient refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Flap Survival Rate | "From enrollment to the end of treatment at 8 weeks"
  The percentage of flaps that survive completely without necrosis or partial loss. Complications will be graded (e.g., total flap loss, partial necrosis, or marginal necrosis).
  Unit: Percentage. Measurement Tool: ruler/(Mesure).

SECONDARY OUTCOMES:
Range of Motion in Reconstructed Area | "From enrollment to the end of treatment at 8 weeks"
  Assessment of the range of motion in the reconstructed area. Unit: Degrees. Measurement Tool: Goniometer.
Strength in Reconstructed Area | "From enrollment to the end of treatment at 8 weeks"
  Evaluation of muscle strength in the reconstructed area. Unit: Newton (N). Measurement Tool: Dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided